CLINICAL TRIAL: NCT04911764
Title: Ability of the 3-minute Step Test Protocol for Detecting Exercise Desaturation Episodes in Chronic Respiratory Insufficiency: Protocol STEPSAT: Three-min Step Test and Exercise Desaturation Detection in Chronic Respiratory Insufficiency Patients
Brief Title: Three-min Step Test and Exercise Desaturation Detection in Chronic Respiratory Insufficiency Patients
Acronym: STEPSAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI19-0003_STEPSAT
Record Dates: First submitted 2021-05-20; First posted 2021-06-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: COPD; Chronic Respiratory Disease
Keywords: COPD; Exercise; oxygen desaturation; field tests
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized interventional study, with low risks and constraints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-min Step Test and Exercise desaturation detection in COPD (Experimental): Each patient recruited will performed both field tests, being therefore his or her own witness.
  Interventions: Diagnostic Test: Three-min Step Test and Exercise desaturation detection in COPD

INTERVENTIONS:
Diagnostic Test: Three-min Step Test and Exercise desaturation detection in COPD — For this research, 2 visits will be scheduled (V1 and V2) for each patient. During V1, after collecting the filled and signed consent form from the patient, anthropometric measurements and pulmonary function assessment will be performed before the realization of a maximal graded test. This inclusion visit will be carried out as part of an inclusion within a respiratory rehabilitation program. During V2, each patient will randomly perform a 6-minute walking test and a 3-minute step test, in similar standard conditions. A 30-minute resting period will be allowed between the two field tests. During the realization of the tests, cardio-respiratory adaptations will be monitored throughout both tests with portable gas analyzer and pulsed oxymetry system.

SUMMARY:
The study project will aim at the evaluation of the occurrence of exercise desaturation phenomenon during two different modalities of exercise (walking and stepping condition). This study will allow determining the sensibility of the 3-minute step test to detect exercise desaturation, in comparison with the gold standard (6-minute walking test). The 3-minute step test could therefore appear as a complementary tool for the evaluation of oxygen desaturation in chronic respiratory disease.

DETAILED DESCRIPTION:
The 6-minute walking test is currently the gold standard for the evaluation of oxygen desaturation phenomenon during exercise and for the adjustment of O2 flow rate. But, due to spatial constraints, this test remains difficult to apply in ecological conditions and the 3-minute step test could be a complementary method to the walking test for the evaluation of chronic respiratory diseases. For this study, patients will perform, during 2 visits, a maximal graded test and two field tests (6-min walking test and 3-min step test) under identical conditions. During these tests, pulsed oxygen saturation and psycho-physiological adaptations to exercise will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged by 18 and more ;
* Patient with an chronic obstructive respiratory insufficiency, confirmed by clinical and functional criteria ;
* Patient with exercise-induced oxygen desaturation ;
* Patient clinical ly stable, with no exacerbation period within the last 2 months before inclusion ;
* Consent form signed by the patient.

Exclusion Criteria:

* Patient in exacerbation period at the inclusion time ;
* Pregnant and breastfeeding women ;
* Patient with orthopedic disorder that could limit the ability of stair climbing;
* Any other disease that could influence exercise capacity of the patient or that could impair exercise test realization ;
* Patient with law protection (guardianship or protection of vulnerable adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Detection of exercise desaturation occurrence | At Visit 2: between Day 3 and Day 15 after Visit 1
  Detection of exercise desaturation occurrence correspond to a fall of SpO2 rest value by at least 4 points during exercise, assessed with the measurement of pulsed oxygen saturation during the different tests.

SECONDARY OUTCOMES:
Patient-perceived sensation of dyspnea | At Visit 2: between Day 3 and Day 15 after Visit 1
  scoring by Borg Category Ratio 10 scale (CR-10)
  * Scale going from 0 to 10
  * 0 being an absence of sensation, 10 a very high sensation or even maximum.
Patient-perceived sensation of lower extremity fatigue | At Visit 2: between Day 3 and Day 15 after Visit 1
  scoring by Borg Category Ratio 10 scale (CR-10)
  * Scale going from 0 to 10
  * 0 being an absence of sensation, 10 a very high sensation or even maximum.
Oxygen consumption (VO2) | At Visit 2: between Day 3 and Day 15 after Visit 1
  This parameter will be obtained from a measuring device (Metamax), allowing a real time measurement and its registration will be collected at the end of the walking and stepping tests.
  Reported value in ml/min/kg : mean value of the last thirty seconds of each test.
CO2 production (VCO2) | At Visit 2: between Day 3 and Day 15 after Visit 1
  This parameter will be obtained from a measuring device (Metamax), allowing a real time measurement and its registration will be collected at the end of the walking and stepping tests.
  Reported value in ml/min/kg : mean value of the last thirty seconds of each test.
Ventilatory output (VE) | At Visit 2: between Day 3 and Day 15 after Visit 1
  This parameter will be obtained from a measuring device (Metamax), allowing a real time measurement and its registration will be collected at the end of the walking and stepping tests.
  Reported value in l/min : mean value of the last thirty seconds of each test.
Heart rate (HR) | At Visit 2: between Day 3 and Day 15 after Visit 1
  This parameter will be obtained from a measuring device (Metamax), allowing a real time measurement and its registration will be collected at the end of the walking and stepping tests.
  Reported value in Beats/min : mean value of the last thirty seconds of each test.
Muscle deoxygenation (delta HHb) | At Visit 2: between Day 3 and Day 15 after Visit 1
  The assessment of muscle deoxygenation observed by near infrared spectroscopy (NIRS) technology.
  Reported value in arbitrary unit : difference between mean HHb value at rest and the lowest HHb value during each exercise

CONTACTS AND LOCATIONS:
Overall Officials: Florent FAVARD, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Chu de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Anthonisen NR. Prognosis in chronic obstructive pulmonary disease: results from multicenter clinical trials. Am Rev Respir Dis. 1989 Sep;140(3 Pt 2):S95-9. doi: 10.1164/ajrccm/140.3_Pt_2.S95. No abstract available. PMID 2675713
- [Background] Barjaktarevic I, Cooper CB. Supplemental Oxygen Therapy for Patients with Chronic Obstructive Pulmonary Disease. Semin Respir Crit Care Med. 2015 Aug;36(4):552-66. doi: 10.1055/s-0035-1556058. Epub 2015 Aug 3. PMID 26238641
- [Background] Borel B, Wilkinson-Maitland CA, Hamilton A, Bourbeau J, Perrault H, Jensen D, Maltais F. Three-minute constant rate step test for detecting exertional dyspnea relief after bronchodilation in COPD. Int J Chron Obstruct Pulmon Dis. 2016 Nov 29;11:2991-3000. doi: 10.2147/COPD.S113113. eCollection 2016. PMID 27942208
- [Background] Borel, B., C. Wilkinson-Maitland, D. Jensen, J. Bourbeau, A. Hamilton, H. Perrault and F. Maltais. Sensitivity of the 3-min step test to detect dyspnea relief following bronchodilation in COPD: a randomized control trial. American journal of respiratory and critical care medicine. 2014;189: A5862.
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Background] Casanova C, Cote C, Marin JM, Pinto-Plata V, de Torres JP, Aguirre-Jaime A, Vassaux C, Celli BR. Distance and oxygen desaturation during the 6-min walk test as predictors of long-term mortality in patients with COPD. Chest. 2008 Oct;134(4):746-752. doi: 10.1378/chest.08-0520. Epub 2008 Jul 14. PMID 18625667
- [Background] Garcia-Talavera I, Tauroni A, Trujillo JL, Pitti R, Eiroa L, Aguirre-Jaime A, Sanchez A, Abreu J. Time to desaturation less than one minute predicts the need for long-term home oxygen therapy. Respir Care. 2011 Nov;56(11):1812-7. doi: 10.4187/respcare.01164. Epub 2011 May 20. PMID 21605486
- [Background] Perrault H, Baril J, Henophy S, Rycroft A, Bourbeau J, Maltais F. Paced-walk and step tests to assess exertional dyspnea in COPD. COPD. 2009 Oct;6(5):330-9. doi: 10.1080/15412550903156317. PMID 19863362
- [Background] Poulain M, Durand F, Palomba B, Ceugniet F, Desplan J, Varray A, Prefaut C. 6-minute walk testing is more sensitive than maximal incremental cycle testing for detecting oxygen desaturation in patients with COPD. Chest. 2003 May;123(5):1401-7. doi: 10.1378/chest.123.5.1401. PMID 12740254
- [Background] Takigawa N, Tada A, Soda R, Date H, Yamashita M, Endo S, Takahashi S, Kawata N, Shibayama T, Hamada N, Sakaguchi M, Hirano A, Kimura G, Okada C, Takahashi K. Distance and oxygen desaturation in 6-min walk test predict prognosis in COPD patients. Respir Med. 2007 Mar;101(3):561-7. doi: 10.1016/j.rmed.2006.06.017. Epub 2006 Aug 8. PMID 16899358